CLINICAL TRIAL: NCT03682965
Title: Texan Allergy & Sinus Center Mountain Cedar Intra-Lymphatic Immunotherapy Study
Acronym: TX-SMILE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Christopher Thompson, MD (Other)
Responsible Party: Sponsor-Investigator, Christopher Thompson, MD, Principal Investigator, Texan Allergy & Sinus Center
Organization: Texan Allergy & Sinus Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TASC-ILIT-MC-2018
Record Dates: First submitted 2018-09-12; First posted 2018-09-25 (Actual); Results first posted 2021-02-26 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-03

CONDITIONS: Allergic Rhinitis Due to Tree Pollen; Allergic Conjunctivitis; Allergic Rhinoconjunctivitis
Keywords: Mountain Cedar; Juniperus Ashei; Pollinosis; Intra-lymphatic
MeSH Terms: conditions — Conjunctivitis, Allergic; Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intra-lymphatic allergenic extract (Experimental): A series of three injections of 0.1 mL (about 2 drops) of the allergenic extract of Mountain Cedar Pollen given every four weeks into a superficial inguinal lymph node through guidance via ultrasonography using a 1-mL hypodermic syringe with a 25-gauge or smaller needle.
  Interventions: Biological: Intra-lymphatic allergenic extract
- Intra-lymphatic placebo (Placebo Comparator): Diluent as placebo control (sterile saline solution containing 0.4% phenol as a preservative and matched concentration of glycerin) given as a series of three injections of 0.1 mL (about 2 drops) every four weeks into a superficial inguinal lymph node through guidance via ultrasonography using a 1-mL hypodermic syringe with a 25-gauge or smaller needle.
  Interventions: Biological: Intra-lymphatic placebo

INTERVENTIONS:
Biological: Intra-lymphatic allergenic extract — Mountain Cedar pollen allergenic extract is an FDA-approved, commercially available product for diagnosis and hypo-sensitization treatment of allergies. The labeled use is deep subcutaneous or percutaneous injection. Hyposensitization treatment is typically a series of 30 - 70 injections over 3 - 5 years into the upper aspect of the arm. This investigation is a proof-of-concept study to evaluate an alternative hyposensitization regimen of 3 injections directly into an inguinal lymph node.
  Other Names: NDC02686614
  Arms: Intra-lymphatic allergenic extract
Biological: Intra-lymphatic placebo — The control group will receive a regimen of 3 injections of diluent (placebo) directly into an inguinal lymph node on the same schedule as the active treatment group.
  Arms: Intra-lymphatic placebo

SUMMARY:
TX-SMILE is an investigator-initiated, multi-center, randomized, double-blind, parallel-group, placebo-controlled study to evaluate the efficacy, safety, and tolerability of intra-lymphatic administration of an approved allergenic extract for the immunotherapy treatment of allergic rhinitis and conjunctivitis due to pollen from the conifer Mountain Cedar.

DETAILED DESCRIPTION:
TX-SMILE is an investigator-initiated, multi-center, randomized, double-blind, parallel-group, placebo-controlled study to evaluate the efficacy, safety, and tolerability of an alternative injection site and associated adjustments to dosing and treatment regimen for allergen immunotherapy with a commercially-available, FDA-approved allergenic extract for the immunotherapy treatment of allergic rhinitis and conjunctivitis due to pollen from the conifer Mountain Cedar (Juniperus ashei).

The purpose of this study is to evaluate the effect of a three-dose treatment series of ultrasonography-guided, intra-lymphatic immunotherapy injections over a two-month period prior to the start of the 2018-2019 Mountain Cedar allergy season in central Texas. Patients will be evaluated for safety and tolerability during the treatment period and for efficacy during the 2018-2019 Texas Mountain Cedar pollen season.

ELIGIBILITY:
Inclusion Criteria:

1. Both male and female adult patients with a history of Season Allergic Rhinitis (SAR) with bothersome symptoms due to Mountain Cedar pollinosis confirmed using the Modified Quantitate Test (MQT; defined as a wheal greater than or equal to 3 millimeters larger than the diluent control)
2. Patients must be willing to provide written, informed consent
3. Patients must be willing and able to comply with study procedures
4. Women of childbearing potential must agree to use an acceptable form of contraception during the trial

Exclusion Criteria:

1. Patients less than 18 years of age
2. Clinically-significant chronic sinusitis, as determined by the investigator
3. History of anaphylaxis during Mountain Cedar skin prick testing
4. Participation in another clinical trial or use of an experimental medication within 30 days of enrollment
5. Medically significant co-morbidities that, in the opinion of the investigator, place the subject at increased risk during the study, including but not limited to:

   1. Autoimmune diseases, other than allergic rhinitis (AR), stable allergic asthma, eczema and food sensitivities
   2. Pulmonary or respiratory diseases other than stable asthma
   3. Cancer other than basal cell carcinoma
   4. Coronary artery disease or hypertension treated with beta-blockers
   5. Clinically significant impairment of renal or hepatic function
6. Use of concomitant medications that, in the opinion of the investigator, may reduce the effectiveness of rescue treatments for anaphylaxis (e.g. beta-blockers) or alter the immune response to allergen immunotherapy (e.g., immunosuppressants, systemic corticosteroids)
7. Previously completed immunotherapy for Mountain Cedar pollinosis, that in the opinion of the investigator would interfere with the assessment or treatment of the patient
8. Inability to access suitable lymph nodes for intralympahtic injections
9. Plans to leave the area for a significant period of the upcoming Mountain Cedar pollen season
10. Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Thompson, MD, Principal Investigator — Texan Allergy & Sinus Center
Locations (3):
- United States (3):
  - Texan Allergy & Sinus Center, Austin, Texas
  - Texan Allergy & Sinus Center, Grapevine, Texas
  - Texan Allergy & Sinus Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thompson CP, Silvers S, Shapiro MA. Intralymphatic immunotherapy for mountain cedar pollinosis: A randomized, double-blind, placebo-controlled trial. Ann Allergy Asthma Immunol. 2020 Sep;125(3):311-318.e2. doi: 10.1016/j.anai.2020.04.030. Epub 2020 May 11. PMID 32407947

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intra-lymphatic Allergenic Extract | Intra-lymphatic Placebo
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intra-lymphatic Allergenic Extract | Intra-lymphatic Placebo | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 34 [25 to 65] | 32 [20 to 57] | 33 [20 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Average Daily Total Combined Score (TCS)
Description: The TCS is the preferred endpoint for rhinoconjunctivitis as recommended by the European Academy of Allergy and Clinical Immunology. Scoring of the TCS is from 0 to 38 on each day that it is assessed. The TCS is the sum of the symptom scores for "runny nose", "stuff nose", "sneezing", "itchy nose", "gritty/itchy eyes", and "watery eyes" rated from no symptoms = 0 to severe symptoms = 3 plus the score for use of rescue medications for allergy symptoms 6 points for oral antihistamine, 6 points for eye drops, and 8 points for a nasal corticosteroid. Thus, a lower score represents fewer symptoms and associated need for allergy medication, while a higher score reflects more severe symptoms and the use of medication to treat symptoms. The TCS will be measured during the 2018-2019 Mountain Cedar pollen se
Time Frame: Up to 4 months
Population: Safety analysis included all participants who received at least one dose of study intervention. Efficacy analyses were on the per protocol dataset, which included participants who received three study treatment injections and completed at least 50% of expected electronic diary responses during the allergy season, with no major protocol violations. aLL enrolled patients met the criteria for inclusion in both the safety and per protocol analysis populations
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intra-lymphatic Allergenic Extract | Intra-lymphatic Placebo
Number analyzed (Participants) | 11 | 10
units on a scale | 10.1 (3.3) | 13.0 (7.8)
Statistical Analysis 1: Comparison: Intra-lymphatic Allergenic Extract vs Intra-lymphatic Placebo; Test type: Superiority; p = 0.004, Kruskal-Wallis

2. Secondary Outcome: Number of Peak Pollen Season Days With a Lower Group Average Total Combined Score
Description: Evaluated during the 2018-2019 Texas Mountain Cedar allergy season. The number of days with a lower group average Total Combined Score, comparatively, in each Arm/Group are reported. Scoring of the TCS is from 0 to 38 on each day that it is assessed.The TCS is the sum of the symptom scores for "runny nose", "stuff nose", "sneezing", "itchy nose", "gritty/itchy eyes", and "watery eyes" rated from no symptoms = 0 to severe symptoms = 3 plus the score for use of rescue medications for allergy symptoms 6 points for oral antihistamine, 6 points for eye drops, and 8 points for a nasal corticosteroid. Thus, a lower score represents fewer symptoms and associated need for allergy medication, while a higher score reflects more severe symptoms and the use of medication to treat symptoms.
Time Frame: Assessed up to 4 months, number of actual peak pollen season days was 27
Measure: Number; unit: days
Arm/Group | Intra-lymphatic Allergenic Extract | Intra-lymphatic Placebo
Number analyzed (Participants) | 11 | 10
days | 20 | 7
Statistical Analysis 1: Comparison: Intra-lymphatic Allergenic Extract vs Intra-lymphatic Placebo; The secondary efficacy endpoint was the percentage of days during peak pollen season for which the average total combined score was lower in the immunotherapy group than in the placebo group; Test type: Superiority; p < 0.05, Clopper-Pearson binomial exact test — The Holm-Bonferroni correction for multiple tests was used because the two outcomes are based on correlated data

3. Secondary Outcome: Patient Reported Pain or Discomfort Following Intra-lymphatic Injections
Description: Patient reported pain will be measured immediately after ILIT procedure using the Numeric Rating Scale 11 (NRS-11 rating scale). The NRS-11 asks patients to rate their pain on a scale from 0 (no pain or discomfort) to 11 (worst possible pain).
Time Frame: Immediately after the ILIT procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intra-lymphatic Allergenic Extract | Intra-lymphatic Placebo
Number analyzed (Participants) | 11 | 10
units on a scale | 0.5 (0.5) | 0.5 (0.5)

4. Secondary Outcome: Patient-reported Treatment Satisfaction at the End of Study
Description: Percentage of patients reporting satisfaction with their treatment
Time Frame: Up to 4 months
Measure: Number; unit: percentage of participants
Arm/Group | Intra-lymphatic Allergenic Extract | Intra-lymphatic Placebo
Number analyzed (Participants) | 11 | 10
percentage of participants | 91 | 90
Statistical Analysis 1: Comparison: Intra-lymphatic Allergenic Extract vs Intra-lymphatic Placebo; Test type: Superiority; p = 0.23, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Percentage Change in Allergen-specific Serum IgE
Description: Percentage change in allergen-specific serum IgE from baseline to the end-of-study visit between active ILIT and placebo.
Time Frame: Assessed prior to the first injection and to 4-8 weeks after the end of the 2018-2019 pollen season
Measure: Mean (Standard Deviation); unit: percentage change in serum IgE
Arm/Group | Intra-lymphatic Allergenic Extract | Intra-lymphatic Placebo
Number analyzed (Participants) | 11 | 10
percentage change in serum IgE | 148 (214) | 201 (231)

6. Secondary Outcome: Total Safety Score (TSS) for Active and Placebo Treatment Groups
Description: The total safety score is a is based on World Allergy Organization grading for allergic reactions. Following allergen or placebo exposure via intra-lymphatic injection, patients are monitored for local and systemic allergic reactions for up to 60 minutes post-procedure. At each exposure, a score is rated on a scale from none = 0, local reactions only = 1, mild systemic reactions (WAO Grade 1/2) = 2, moderate systemic reaction (WAO Grade 3) = 3, and severe systemic reaction (WAO grade 4) = 4. The total safety score for each group is the sum of the individual scores of each patient across all three treatments (exposures). Thus, the subject may have a score from 0 to 12 with 0 reflecting no allergic reaction to the allergen and 12 reflecting severe allergic reactions, and the TSS for a group is the sum for all patients in the group. The TSS is used to elicit and grade adverse events of interest rather than for statistical analysis.
Time Frame: 8 weeks
Measure: Number; unit: score on a scale
Arm/Group | Intra-lymphatic Allergenic Extract | Intra-lymphatic Placebo
Number analyzed (Participants) | 11 | 10
score on a scale | 3 | 1

7. Secondary Outcome: Number of Subjects Who: Experienced Anaphylaxis, Were Treated With Epinephrine, or Experienced Any Other Treatment-emergent SAE Within 60 Minutes of Any of Three Planned ILIT Procedures
Description: To evaluate the safety of ILIT for Mountain Cedar pollinosis relative to placebo control based on the proportion of subjects receiving allergenic extract versus the proportion of subjects receiving placebo that:
  1. experience anaphylaxis, or
  2. are treated with epinephrine, or
  3. experience any other treatment-emergent, serious adverse event (SAE) within 60 minutes of any of the three planned ILIT procedures.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intra-lymphatic Allergenic Extract | Intra-lymphatic Placebo
Number analyzed (Participants) | 11 | 10
Participants | 0 | 0

8. Other Pre Specified Outcome: Total Number of Rescue Inhaler Uses by Patients With Asthma
Description: Relative use of rescue inhalers by patients with comorbid asthma between active and placebo groups during the 2018-2019 Mountain Cedar pollen season.
Time Frame: Up to 4 month
Measure: Number; unit: Rescue Inhaler Uses
Arm/Group | Intra-lymphatic Allergenic Extract | Intra-lymphatic Placebo
Number analyzed (Participants) | 11 | 10
Rescue Inhaler Uses | 0 | 0

ADVERSE EVENTS:
Time Frame: From the start of treatment (1st ILIT injection) through the end of the pollen season and for two months therafter, an average of 4 months per participant.
Description: In addition to spontaneous reporting and safety monitoring procedures, including vital signs assessments, Adverse Events of Interest were collected using the Total Safety Score worksheet during each injection procedure.
Arm/Group | Intra-lymphatic Allergenic Extract | Intra-lymphatic Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 5/11 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intra-lymphatic Allergenic Extract (N=11) | Intra-lymphatic Placebo (N=10)
Injection-site redness (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Injection-site bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
hypertension (Cardiac disorders) | 1 (1) | 0 (0) — transient elevation in blood pressure during post-injection monitoring
peri-procedural anxiety (General disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/65/NCT03682965/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT03682965/SAP_001.pdf
  • Informed Consent Form (2018-12-24): https://cdn.clinicaltrials.gov/large-docs/65/NCT03682965/ICF_002.pdf